CLINICAL TRIAL: NCT04037878
Title: Opioid Consumption Following TAP Block Versus Intraperitoneal/Incisional Bupivicaine in Patients Undergoing Major Gynecologic Surgeries: A Randomized Controlled Trial
Brief Title: Tap Block vs Peritoneal Infiltration After Major Gynecological Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Samina Ismail, Professor of Anesthesiology, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AgaKhan1
Record Dates: First submitted 2019-06-20; First posted 2019-07-30 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Pain, Acute
Keywords: TAP block; Local infiltration; Tramadol; Gynecological surgery; Pain control
MeSH Terms: conditions — Acute Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The patient is randomized according to randomization block and sealed envelops. The investigator doesn't know what study group the patient is randomized into
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- TAP block group (Experimental): Patients in this arm will be given Transversus Abdominal Plane(TAP) block after the induction of anesthesia. They will also be given post operative patient controlled intravenous analgesia(PCIA) using tramadol.
  Interventions: Procedure: Transversus Abdominis Plane Block(TAP Block); Drug: PCIA Tramadol
- Local infiltration (Experimental): Patients in this arm will be given local and intraperitoneal infiltration of local anesthetic before closure.They will also be given post operative patient controlled intravenous analgesia(PCIA) using tramadol.
  Interventions: Procedure: Intra-peritoneal infiltration; Drug: PCIA Tramadol
- Control group (Other): These patients will be given post operative analgesia in the form of patient controlled intravenous analgesia(PCIA) using tramadol. Neither local infiltration nor TAP block will be administered
  Interventions: Drug: PCIA Tramadol

INTERVENTIONS:
Procedure: Transversus Abdominis Plane Block(TAP Block) — Under ultrasound guidance, a 22 gauge stimuplex needle will be used to approach the transversus abdominis plane and 20ml of 0.25% Bupivicaine will be infiltrated into the TAP space. This procedure will be performed on either sides once anesthesia is induced.
  Arms: TAP block group
Procedure: Intra-peritoneal infiltration — Before skin closure, the surgeon will infiltrate the peritoneal cavity using a mixture of bupivicaine and epinephrine
  Arms: Local infiltration
Drug: PCIA Tramadol — All patients will be given patient controlled intravenous analgesia using Tramadol as the drug

SUMMARY:
It is a randomized controlled trial to determine the total tramadol consumption after major gynecological studies. Intervention groups include TAP block or local infiltration by the surgeon. These will be compared to a control group. Total tramadol consumption will be calculated and therefore pain control will be assessed.

DETAILED DESCRIPTION:
All patients will receive standardized general anesthetic with standard monitoring. Anesthesia will be induced with intravenous (IV) tramadol (1milligram/kg), propofol (2 mg/kg) and atracurium 0.5mg/kg. Anaesthesia will be maintained with oxygen/air (40:60) with one MAC(Minimum Alveolar Concentration) of isoflurane.

TAP block will be performed for Group T patients before surgical incision with the help of an ultrasound and will be performed by two of the anesthesiologists who are part of this study. The study drug for the TAP block will be two syringes of 20 ml containing bupivacaine 0.25% with no other additives. For the infiltration group I, a 50ml syringe will contain 25ml of 0.5% Bupivacaine and 25ml of 5mics/ml epinephrine. These solutions will be made there and then by the anesthesiologist and the drugs for these solutions will be provided by the clinical trial unit. Allocation to group T, I and C will be according to the randomization block explained earlier. For group T, the US-guided TAP block technique will be similar to the method described by Hebbard and colleagues; (21) an ultrasound linear probe will be positioned in the mid-axillary line in the axial plane half-way between the iliac crest and the costal margin. Transversus abdominal plain will be located under ultrasound guidance. One ml test injection of the study solution will be permitted to confirm needle location. A total of 20ml of study solution will be injected on each side after aspiration to avoid intravascular placement. Surgical incision will be given after 20 minutes of TAP. Additional doses of Tramadol 10mg IV stat will be given on need basis (Rise of heart rate and blood pressure more than 20 % of baseline).

Towards the end of surgery, 50 ml of solution prepared by the anesthesiologist will be used for Group I. 50ml of 0.25% Bupivicaine with epinephrine will be poured into a sterile galley pot, from which the surgeon will draw up the solution. The surgeon will be asked to spray 10ml of this solution on to the pouch of Douglas, 10ml in the peritoneum, 10ml in the rectus sheath and 20ml in the skin.

The amount of Bupivicaine used for group I and T is less than the maximum safe dose which is 2.5mg per kg. Minimal side effects are reported using an ultrasound guided TAP block technique(22). If an immediate side effect is noted while performing the technique, treatment will be administered and the patient will be withdrawn from the study.

The control group (C) will receive the standard anesthesia and analgesia as mentioned above without any nerve block technique.

Prophylactic antiemetics in the form of ondansetron 4mg IV stat block and IV paracetamol 15mg/kg will be administered 30 minutes before the end of surgery and diclofenac 100 mg suppository will be administered at the end of surgery.

Routine monitoring of intraoperative blood pressures, heart rates, (base line, induction, surgical incision and at 10 minutes interval) administered fluid and drugs, surgical time and estimated blood loss will be recorded on intraoperative chart.

After completion of the surgical procedure, patients will be transferred to the post anesthesia care unit (PACU). A standardized postoperative analgesic regimen, consisting of regular rectal diclofenac 100 mg every 12 hours and oral paracetamol 1000mg every 6 hrs combined with IV PCIA Tramadol (no baseline infusion, demand bolus dose 15 mg, lock out 8 min), will be commenced on admission to the PACU for all 3 groups. Total tramadol consumption and side effects will be calculated at end of 12 hours.

ELIGIBILITY:
Inclusion Criteria:

* Weight between 40 and 90kg
* ASA(American Society of Anesthesiologists) I to III
* Females scheduled for major gynecological surgeries(Abdominal hysterectomy, myomectomy, ovarian cystectomy, oophorectomy) through Pfannenstiel incision

Exclusion Criteria:

* Refusal to participate in the study,
* History of drug allergy to bupivacaine, tramadol or other narcotics, addiction/ tolerance to opioids,
* Having bleeding disorders,
* Abdominal skin infections or open wounds/ abdominal drains,
* Previous history of failed TAP block,
* On blood thinners or narcotic analgesia

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2020-06-23 (Actual); Study Completion 2020-06-23 (Actual)

PRIMARY OUTCOMES:
Total consumption of tramadol | 12 hours post operatively
  Total consumption of tramadol post operatively

SECONDARY OUTCOMES:
Pain score | 12 hours post operatively
  Will be measured on a numerical rating scale which will be between 0-10
Respiratory depression | 12 hours post operatively
  Less than 10 breaths per minute would be considered as respiratory depression
Nausea | 12 hours post operatively
  Nausea and vomiting will be measured by verbal descriptive scale between 0-3
Sedation | 12 hours post operatively
  Will be measured according to the following 0 Awake / alert. 1 Sleepy / responds appropriately. 2 Somnolent / arousable (light stimuli). 3 Deep sleep / rousable (deeper physical stimuli)
Patient satisfaction | 12 hours post operatively
  7-point Likert scale (1=strongly disagree, 7=strong¬ly agree). Total satisfaction score was calculated from sum of response

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan Hospital, Karachi, Sindh, Pakistan

REFERENCES:
- [Background] Size M, Soyannwo OA, Justins DM. Pain management in developing countries. Anaesthesia. 2007 Dec;62 Suppl 1:38-43. doi: 10.1111/j.1365-2044.2007.05296.x. PMID 17937712
- [Result] Stanley G, Appadu B, Mead M, Rowbotham DJ. Dose requirements, efficacy and side effects of morphine and pethidine delivered by patient-controlled analgesia after gynaecological surgery. Br J Anaesth. 1996 Apr;76(4):484-6. doi: 10.1093/bja/76.4.484. PMID 8652316